CLINICAL TRIAL: NCT06797466
Title: Investigation of the Effect of Three Dimensional Virtual Reconstruction (3D) on Percutaneous Nephrolithotomy Learning Curve in Specialist Training
Brief Title: Three Dimensional Virtual Reconstruction (3D) in Percutaneous Nephrolithotomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University (Other)
Responsible Party: Principal Investigator, Bedreddin Kalyenci, Principal Investigator, Adiyaman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HRÜ/24.21.44
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-01

CONDITIONS: PNL; Stone, Kidney
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3D imaging technique on the PCNL (Experimental)
  Interventions: Procedure: 3D imaging technique on the PCNL
- standard PCNL (No Intervention)

INTERVENTIONS:
Procedure: 3D imaging technique on the PCNL — Establishing a percutaneous access route for the stone is the first and most important step in PCNL surgery. Choosing the perfect route, position and direction largely depends on surgical experience and the ability to understand renal/peri-renal anatomy. In general, a good CT scan of the abdomen and pelvis and an experienced surgeon are sufficient, but this requires significant time in the learning curve. The aim of our study is to investigate the effect of 3D imaging technique on the PCNL learning curve in specialist training.
  Arms: 3D imaging technique on the PCNL

SUMMARY:
The aim of our study is to investigate the effect of 3D imaging technique on the PCNL learning curve in specialist training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with kidney stones larger than 2 cm and those with PCNL indication.

Exclusion Criteria:

* Patients with missing CT images, missing clinical information, or inaccessible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with perioperative Bleeding. | immediately after the intervention/procedure/surgery
Number of Participants with stone free | 1 month after the intervention/procedure/surgery
leng of the hospital stay | immediately after the intervention/procedure/surgery

SECONDARY OUTCOMES:
Number of Participants with Complication | immediately after the intervention/procedure/surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)